CLINICAL TRIAL: NCT03699865
Title: Young Adults and Low Nicotine Cigarettes
Acronym: YLP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa Mercincavage, Research Assistant Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UPCC 10021; 1K07CA218366-01A1 (NIH); 829101 (Other: University of Pennsylvania IRB number)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Smoking
Keywords: low nicotine; smoking behaviors; risk perceptions
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, 2 x 4 mixed factorial design laboratory-based study manipulating: (1) cigarette pack color (4-level within-subjects factor: own brand vs. white vs. purple vs. black color), and (2) nicotine content (2-level between-subjects factor: moderate vs. very low nicotine content). All participants will provide and smoke their preferred brand for an initial 5-day baseline period, receiver their own brand free-of-charge for 5-days, and then will be randomly assigned to smoke either intermediate or very low LNC cigarettes for the study duration. We will supply participants with LNC cigarettes in three pack colors; each color will be used for a 10-day period, in counter-balanced order.
Who Masked: Participant
Masking Description: Participants will be informed that they will be supplied cigarettes with low nicotine content but will be blinded to exact nicotine content and unaware that within-subject, all packages will contain the same type of low nicotine cigarette
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Purple (Experimental): Participants will receive cigarettes with intermediate or very low nicotine content in purple packaging
  Interventions: Other: Nicotine content
- White (Experimental): Participants will receive cigarettes with intermediate or very low nicotine content in white packaging
  Interventions: Other: Nicotine content
- Black (Experimental): Participants will receive cigarettes with intermediate or very low nicotine content in black packaging
  Interventions: Other: Nicotine content

INTERVENTIONS:
Other: Nicotine content — Study-supplied cigarettes will contain either intermediate or very low nicotine content

SUMMARY:
The purpose of this study is to look at the effects of investigational low nicotine cigarettes on young adult smokers. The investigators are interested in how using these products affects young adults' perceptions and smoking behaviors. This research may help inform the Food and Drug Administration (FDA) how best to regulate tobacco products in the future with the goal of improving public health.

DETAILED DESCRIPTION:
Investigators will recruit 100 young adult cigarette smokers to a 40-day, laboratory-based protocol. You will provide and smoke your preferred brand cigarettes for an initial 5-day baseline period, then receive your own brand free-of-charge for an additional 5-day period, and then will receive free, investigational low nicotine cigarettes for the remaining study duration (i.e., 30 days total). Low nicotine cigarettes will be provided in three varieties; each variety will be used for a 10-day period, in counterbalanced order. Primary outcomes will include smoking behaviors (daily cigarette consumption and total puff volume), harm perceptions (i.e., beliefs about product safety), and tobacco exposure (i.e., carbon monoxide [CO]). You will complete in-person visits at the Center for Interdisciplinary Research on Nicotine Addiction (CIRNA) every 5 days, for a total of nine in-person visits.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be 100 male and female young adult smokers who:

  * Are aged 18-25
  * Report smoking ≥ 100 lifetime cigarettes
  * Report smoking at least 1 non-menthol, filtered cigarette per day

Exclusion Criteria:

* We will exclude those who:

  * Plan to quit smoking in the next month
  * Smoke menthol cigarettes > 80% of the time
  * Report consuming ≥ 25 alcohol-containing drinks per week
  * Report a history or current psychiatric diagnosis or severe medical condition,
  * Are color-blind or have another visual impairment (e.g., partial blindness, uncorrected cataract)
  * Are pregnant and/or lactating

Additional, general reasons for exclusion include:

* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible at any point throughout the study.
* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
* Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Daily cigarette consumption | Days 0 through 40
  Daily cigarette consumption will be assessed primarily by participant self-report and secondarily through collection of spent filters for all cigarettes smoked during the 35-day study period, and will be averaged across baseline and pack color periods.

SECONDARY OUTCOMES:
Total puff volume | Days 0, 5, 10, 15, 20, 25, 30, 35, and 40
  Total puff volume (total smoke inhaled per cigarette) will be collected twice during laboratory visits using a handheld, portable, electronic topography device. Assessments will be averaged across study periods.
Risk perceptions | Days 10, 20, 30, and 40
  Perceptions of risks of using study cigarettes will be assessed at the end of own brand and pack color periods using individual items and a summary score from an 8-item, 5-point Likert scale (1 = "definitely untrue", 5 = "definitely true") stating: "Compared to your own cigarettes, the cigarettes you are currently smoking…": a) "are lower in nicotine", b) "are lower in tar", c) "are less addictive", d) "are less likely to cause cancer", e) "have fewer chemicals", f) "are healthier", g) "make smoking safer", h) "help people quit smoking."
Harm exposure | Days 0, 5, 10, 15, 20, 25, 30, 35, and 40
  Harm exposure will be approximated by changes in expired air carbon monoxide (CO), a commonly used biochemical measure of tobacco smoke exposure that is sensitive to changes in puffing behavior. We will assess CO at the onset of each visit to represent daily exposure, as well as before and after each cigarette smoked during laboratory visits. The change in CO values resulting from smoking a cigarette will estimates smoke exposure due to smoking an individual cigarette.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Mercincavage, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided